CLINICAL TRIAL: NCT03607968
Title: Factors Affecting the Improvement of Severity of Concomitant Urodynamic Stress Incontinence After a Novel Transvaginal Mesh Surgery for Women With Pelvic Organ Prolapse
Brief Title: Factors Affecting the Improvement of Severity of Concomitant USI After a Novel TVM Surgery for Women With POP
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201604022RIND
Record Dates: First submitted 2018-05-13; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2016-05

CONDITIONS: Concomitant Conditions
Keywords: Pelvic organ prolapse; Transvaginal mesh; Urodynamic stress incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All women in this study: All women with POP and concomitant overt or occult USI, who underwent the novel anterior TVM surgeries, were enrolled in this study. Medical records, including urodynamic studies, questionnaires and 3-day bladder diaries, were retrospectively reviewed. Linear regress analysis was used to identify factors that were responsible for the changes in pad weights from baseline [i.e., 100 * (postoperative pad weight - baseline pad weight)/baseline pad weight].
  Interventions: Procedure: The novel anterior TVM surgeries

INTERVENTIONS:
Procedure: The novel anterior TVM surgeries — A novel transvaginal mesh (TVM) surgery fro women with pelvic organ prolapse (POP) had been reported. Chang TC, Hsiao SM, Chen CH, Wu WY, Lin HH. Clinical outcomes and urodynamic effects of tailored transvaginal mesh surgery for pelvic organ prolapse. Biomed Res Int http;//dx.doi.org/10.1155/2015/191258.

SUMMARY:
Background/Purpose:

A novel transvaginal mesh (TVM) surgery for women with pelvic organ prolapse (POP) had been reported. However, factors affecting the efficacy of this novel TVM surgery are unknown; and the above information should be important for preoperative consultation, especially for POP women with concomitant urodynamic stress incontinence (USI). Thus, the aim of this study is to investigate the factors responsible for anti-incontinence effect of this novel anterior TVM surgery.

Patients and Methods:

All women with POP and concomitant overt or occult USI, who underwent the novel anterior TVM surgeries, were enrolled in this study. Medical records, including urodynamic studies, questionnaires and 3-day bladder diaries, were retrospectively reviewed. Linear regress analysis was used to identify factors that were responsible for the changes in pad weights from baseline [i.e., 100 * (postoperative pad weight - baseline pad weight)/baseline pad weight].

Expected Results:

The investigators will get the factors responsible for anti-incontinence effect of this novel anterior TVM surgery. Key Words: pelvic organ prolapse, stress urinary incontinence, pad test, urodynamic stress incontinence

DETAILED DESCRIPTION:
Background/Purpose:

A novel transvaginal mesh (TVM) surgery for women with pelvic organ prolapse (POP) had been reported. However, factors affecting the efficacy of this novel TVM surgery are unknown; and the above information should be important for preoperative consultation, especially for POP women with concomitant urodynamic stress incontinence (USI). Thus, the aim of this study is to investigate the factors responsible for anti-incontinence effect of this novel anterior TVM surgery.

Methods:

All women with POP and concomitant overt or occult USI, who underwent the novel anterior TVM surgeries between November 2011 and December 2015 at the Department of Obstetrics & Gynecology, were enrolled in this study. Medical records, including urodynamic studies, questionnaires and 3-day bladder diaries, were retrospectively reviewed. Linear regress analysis was used to identify factors that were responsible for the changes in pad weights from baseline [i.e., 100 * (postoperative pad weight - baseline pad weight)/baseline pad weight].

Expected Results:

The investigators will get the factors responsible for anti-incontinence effect of this novel anterior TVM surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosed with pelvic organ prolapse and concomitant overt or occult urodynamic stress incontinence
* Received the novel anterior transvaginal mesh surgery.

Exclusion Criteria:

* Pregnant women, prepare for pregnancy or younger than 20-year-old
* Significant severe urinary urgency
* Mixed urinary incontinence with dominant urgency incontinence
* Regular urethral catheterization or intermittent self-catheterization
* Urinary tract infection (UTI) or chronic inflammation in recent 2 weeks before operation
* Bladder calculus
* A history of pelvic radiotherapy
* Preexisting malignant pelvic tumors.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women with POP and concomitant overt or occult USI, who underwent the novel anterior TVM surgeries, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of urodynamic stress incontinence | 2011/11/01-2015/12/31
  Preoperative and postoperative urodynamic studies to detect USI

SECONDARY OUTCOMES:
Improvement of stress urinary incontinence | 2011/11/01-2015/12/31
  Preoperative and postoperative 20-minute pad test changes

CONTACTS AND LOCATIONS:
Overall Officials: HO-HSIUNG LIN, Professor, Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University College of Medicine and Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan